CLINICAL TRIAL: NCT06408844
Title: The Effects of Physical Activity Behavior Change Program Implemented With 5A Model on Physical and Psychosocial Health in School Age Children
Brief Title: Examining the Impact of Behavior Change Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Filiz Özdemir, associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Inonu-FTR-MHK-01
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Physical Inactivity; Behavior, Health; Health Behavior
Keywords: 5A Model; child; behaviour change; physical activity; health promotion
MeSH Terms: conditions — Sedentary Behavior; Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: There are two groups in this study: the experimental group and the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Training to improve physical activity behavior will be given to the experimental group for 8 weeks, based on the 5A model.
  Interventions: Behavioral: Physical activity behavior change program implemented with 5A model
- Control group (No Intervention): The control group will not receive any intervention and will be asked to continue their routine lives.

INTERVENTIONS:
Behavioral: Physical activity behavior change program implemented with 5A model — According to the 5A model, the personal action plan includes the following items:
  1. List specific goals by behavioral period
  2. List obstacles and strategies to address them
  3. Determine follow-up plan
  4. Sharing the plan with the child and family In accordance with this plan, it is aimed to increase physical activity behavior in the classroom and during online meetings for 8 weeks. Additionally, after the training, motivational reminders will be held at regular intervals until the 28th week.
  Arms: Experimental group

SUMMARY:
The health-related benefits of physical activity are well established for all age groups. It also has positive effects on memory, executive function and school performance in children and adolescents. However, it is known that 81% of individuals between the ages of 11-17 live a life that is not physically active enough. The World Health Organization recommends interventions to increase physical activity. In this study, 48 students from 5th, 6th and 7th grades will be selected from randomly selected secondary schools in Karaman central district and will be divided into experimental and control groups. In this randomized controlled study, behavior change intervention with the 5A model will be applied to the experimental group, and no intervention will be applied to the control group. Physical activity levels, physical and psychosocial health of children in both groups will be evaluated at the beginning of the intervention, at Week 8 and at Week 28. Physical activity diary, "Physical activity scale for 4-8 Grades" scale will be used to measure children's physical activity levels. For their physical health, body composition, strength, flexibility and functional capacity will be evaluated. Quality of life with the "Pediatric Quality of Life 4.0 Inventory" for psychosocial health; Cognitive functions will be evaluated with "CNS Vital Signs Cognitive Performance and Attention Tests". This study aims to evaluate the sustainability effect of the 5A intervention on physical activity and its impact on physical health and psychosocial health.

DETAILED DESCRIPTION:
Behavioral interventions for health promotion are widely used for preventive health practices. There are many studies on topics such as smoking, diet, obesity and oral care. However, we see that studies improving physical activity behavior in children are limited. Considering that physical activity is an important health-related behavior that should be acquired from childhood, we predict that studies on this subject will have an important place in the literature. In addition, it is stated in the guidelines that while the effect of physical activity behavior on health-related parameters in children is clear, more evidence is still needed on its effect on cognitive functions. With our study, we aim to examine the sustainability, physical and psychosocial effects of developing physical activity behavior in children using the 5A model and contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being a middle school student
* Being between the ages of 10-12
* Getting <3.16 points from the "Physical activity scale for grades 4-8"

Exclusion Criteria:

* Having a condition where exercise is contraindicated
* Families or children do not give consent to participate in the study.
* Having a psychosocial problem that prevents adaptation to work

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | 1 day
  Children's physical activity level will be determined using the Paq-c survey.
Physical health | 1 day
  Children's body composition, aerobic capacity, anaerobic capacity, strength and flexibility will be evaluated.
Psychosocial Health | 1 day
  Children's psychosocial health will be assessed with the CNSVS procedure.

SECONDARY OUTCOMES:
Physical Activity attitude | 1 day
  Their attitudes towards Physical Activity will be evaluated.
Behavior Change Step | 1 day
  It will be questioned whether the physical activity behavior is in the pre-contemplation, contemplation, preparation, action or maintenance periods.
Children's Quality of Life | 1 day
  The impact of education on the quality of life will be evaluated using the "Quality of Life Scale for Children".

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Özdemir, Ass. Prof., Principal Investigator — Inonu University
Locations (1):
- Alparslan Ortaokulu, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No